CLINICAL TRIAL: NCT05048186
Title: Refining the Shared Decision Making Process Survey in ADHD Medication Decisions
Status: Completed | Type: Observational
Sponsor: Massachusetts General Hospital (Other)
Collaborators: University of Massachusetts, Boston (Other)
Responsible Party: Principal Investigator, Karen Sepucha, Director of the Health Decision Sciences Center, Massachusetts General Hospital
Other Study IDs: 2019P001434-3
Record Dates: First submitted 2021-03-29; First posted 2021-09-17 (Actual); Results first posted 2024-11-21 (Actual); Last update posted 2024-11-21 (Actual); Status verified 2024-10

CONDITIONS: ADHD
Keywords: shared decision making
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Decision Aid Arm: Participants in this arm will review educational material from the ADHD Decision Aid developed by the Cincinnati Children's Hospital Medical Center.
  Interventions: Behavioral: Attention Deficit Hyperactivity Disorder Treatment Decision Aid
- Control Arm: Participants in this group will not receive any educational materials.

INTERVENTIONS:
Behavioral: Attention Deficit Hyperactivity Disorder Treatment Decision Aid — The parent pre-visit cards from the Cincinnati Children's Hospital's Attention Deficit Hyperactivity Disorder (ADHD) Treatment for School Age Children Decision Aid were used in this study. The 6 pre-visit cards provide an overview of ADHD treatment options, the respective benefits and downsides of each option, and questions to elicit goals/preferences. The four different treatment options presented were: (1) watchful waiting, (2) behavioral treatment, (3) medication treatment, and (4) combined treatment (behavioral and medication together).
  Groups: Decision Aid Arm

SUMMARY:
This is a retrospective observational survey study. We will survey a sample of adult parents or legal guardians who have a child who has been diagnosed with Attention Deficit Hyperactivity Disorder (ADHD) and who discussed ADHD treatment options for their child with a health care provider within the last 2 years. The main goal is to gather evidence of the validity and reliability of the Shared Decision Making Process scale. Secondary goal is to gather evidence on the quality of decisions parents make about their children with ADHD. A third goal is to assess the impact of a Decision Aid on participant knowledge of ADHD treatment options. Participants will be randomized to one of two arms: participants in the intervention arm will review a Decision Aid (patient educational tool) partway through the survey and those in the control arm will not receive any educational materials. All participants will complete survey that includes the Shared Decision Making process survey along with a few other measures. A subset of respondents will also complete a retest survey about two weeks after the initial survey.

DETAILED DESCRIPTION:
This is a retrospective observational survey study. We will survey a sample of adult parents or legal guardians who have a child who has been diagnosed with Attention Deficit Hyperactivity Disorder (ADHD) and who discussed ADHD treatment options for their child with a health care provider within the last 2 years. The main goal is to gather evidence of the validity and reliability of the Shared Decision Making Process scale. Secondary goal is to gather evidence on the quality of decisions parents make about their children with ADHD. A third goal is to assess the impact of a Decision Aid on participant knowledge of ADHD treatment options. Participants will be randomized to one of two arms: participants in the intervention arm will review a Decision Aid (patient educational tool) partway through the survey and those in the control arm will not receive any educational materials. All participants will complete survey that includes the Shared Decision Making process survey along with a few other measures. A subset of respondents will also complete a retest survey about two weeks after the initial survey.

Study staff are working with a national sampling firm to recruit subjects and obtain 500 responses. The sample size was determined to ensure 80% power to detect difference of 0.25SD at 0.05 significant between intervention and control arm on participant knowledge scores. The decision aid intervention consists of a set of pre-visit summary cards for parents that cover the different treatment options and was developed by the Cincinnati Children's Hospital Medical Center.

For the analyses, study staff will examine the descriptives of the Shared Decision Making Process items and knowledge scores for the two arms. Study staff will examine rates of missing data to determine acceptability, and will examine descriptive results to see whether the scores span the range of total possible scores, are normally distributed, and whether there is evidence of floor or ceiling effects. Study staff will also test several hypotheses to examine validity of the scores such as whether higher shared decision making process scores are associated with less decisional conflict and less regret. Staff will also examine retest reliability of the Shared Decision Making Process scale.

ELIGIBILITY:
Inclusion Criteria:

* Adult parent or legal guardian of a child between the ages of 5 and 13 who has been diagnosed with Attention Deficit Hyperactivity Disorder (ADHD)
* Read English
* Have talked with a health care provider about medication for treatment of ADHD for the child in the past 2 years

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Sample was an online non-probability panel of adults living in the United States. Marketing Systems Group, the sample vendor, invited potential respondents from an online panel of adults who had a child with ADHD, and who discussed treatment options for their child's ADHD in the past 2 years.
Sampling Method: Non-Probability Sample
Enrollment: 512 (Actual)
Dates: Start 2021-02-24 (Actual); Primary Completion 2021-03-23 (Actual); Study Completion 2021-04-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Karen Sepucha, PhD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
The study team will create a complete, cleaned, de-identified copy of the final dataset. After the main analyses have been published, information for accessing the data will be made available on the Health Decision Sciences Center website and in publications of the data. Dr. Sepucha will share a de-identified data set with outside investigators at no cost, according to approved Massachusetts General Hospital/Partners policies for data sharing. Investigators from other sites will be able to request the data and will be required to complete a data use agreement that ensures that all local Institutional Review Board requirements are met before using the data, that they will not attempt to identify any data in the dataset, and that they will not share the data set with anyone outside their project team.
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: Data will be available within 3 months after the main results have been published.
Access Criteria: Investigators from other sites will be able to request the data from the principal investigator and will be required to complete a data use agreement that ensures that all local Institutional Review Board requirements are met before using the data, that they will not attempt to identify any data in the dataset, and that they will not share the data set with anyone outside their project team.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Eligible participants were recruited through a national sampling firm, but the sample itself was not a national probability sample. The survey was administered between February 2021 and March 2021. A subset of participants were invited to complete a brief follow-up survey to examine short term test-retest reliability.
Pre-assignment Details: Eligible participants were caregivers who self-identified as having at least one child between the ages of 5 and 13 years old with ADHD and who had talked with a health care provider about starting, stopping, or changing an ADHD medicine in the last 2 years.
Period: Overall Study
Arm/Group | Decision Aid Arm | Control Arm
Started | 252 | 260
Completed | 242 | 256
Not Completed | 10 | 4
Not completed — inconsistent answers for main decision for adhd treatment | 9 | 0
Not completed — did not have sufficient information to calculate the SDM Process score (primary outcome) | 1 | 4

BASELINE CHARACTERISTICS:
Population: Participants provided enough information to calculate the shared decision making process score (primary outcome of interest). Participants were not included in the analytic dataset if they provided inconsistent answers (e.g. indicating their main decision was to start taking medication but they reported their child was not on medication currently and had not been on medication in the past)
Groups:
- Total: Total of all reporting groups
Arm/Group | Decision Aid Arm | Control Arm | Total
Number analyzed (Participants) | 242 | 256 | 498
Age, Continuous [Mean (Standard Deviation); unit: years] — Age of adult caregiver
  years | 37.7 (5.2) | 37.5 (5.8) | 37.6 (5.5)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Female | 166 | 172 | 338
  Male | 75 | 84 | 159
  Unknown | 1 | 0 | 1
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic Only | 20 | 19 | 39
  White, non Hispanic | 168 | 169 | 337
  Black | 30 | 34 | 64
  Asian | 7 | 13 | 20
  Pacific Islander | 0 | 0 | 0
  American Indian | 2 | 2 | 4
  Other | 3 | 6 | 9
  Multiple Races | 10 | 8 | 18
  Unknown | 2 | 5 | 7
Region of Enrollment [Number; unit: participants]
  United States | 242 | 256 | 498

OUTCOME MEASURES:

1. Primary Outcome: Shared Decision Making Process Score
Description: The Shared Decision Making Process scale is a short patient-reported survey that measures the amount of shared decision making that occurs in an interaction. Scores range from 0-4 where higher values indicate a better shared decision making process occurred.
Time Frame: baseline survey (reflecting on the last 24 months)
Population: participants who provided enough information to calculate a shared decision making process score (primary outcome of interest). 498/498 patients provided an answer to this question.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Decision Aid Arm | Control Arm
Number analyzed (Participants) | 242 | 256
units on a scale | 2.83 (1.06) | 2.77 (1.04)
Statistical Analysis 1: Comparison: Decision Aid Arm vs Control Arm; we tested to see whether SDM Process scores were different between patients who received the Decision Aid Arm vs the control arm; Test type: Other; p = 0.503, t-test, 2 sided; Mean Difference (Final Values) = 0.060, 95% CI 2-sided [-0.116 to 0.236]

2. Secondary Outcome: ADHD Knowledge
Description: Multiple choice knowledge items are scored correct/incorrect and a total knowledge score (0-100%) is calculated with higher scores indicating higher knowledge.
Time Frame: baseline survey
Population: participants who completed at least 60% of the knowledge questions. Only 478/498 participants provided sufficient information to calculate a knowledge score.
Measure: Mean (Standard Deviation); unit: percentage of correct answers
Arm/Group | Decision Aid Arm | Control Arm
Number analyzed (Participants) | 239 | 239
percentage of correct answers | 68.37 (22.85) | 59.9 (18.99)

3. Secondary Outcome: Decisional Conflict Tool (SURE)
Description: Measures decisional conflict, consists of 4 yes/no items. Scores range 0-4 where 0 indicates extremely high decisional conflict, 4 indicates no decisional conflict. The number who get score of 4 is reported indicating no decisional conflict. This reports number of participants were reported no decision conflict.
Time Frame: baseline survey
Population: participants who answered all 4 items of the decisional conflict scale. Only 485/498 provided sufficient information to calculate a SURE score.
Measure: Count of Participants; unit: Participants
Arm/Group | Decision Aid Arm | Control Arm
Number analyzed (Participants) | 235 | 250
Participants | 164 | 184

4. Secondary Outcome: Single-item Measure of Decision Regret
Description: Single item asking "If you knew then what you know now, do you think you would make the same decision.
  Response options are:
  Definitely yes, Probably yes, Probably no, Definitely no.
Time Frame: baseline survey
Population: Participants who answered the single-item regret question. Only 497/498 participants provided sufficient information to calculate regret.
Measure: Count of Participants; unit: Participants
Arm/Group | Decision Aid Arm | Control Arm
Number analyzed (Participants) | 242 | 255
Participants
  Definitely Yes | 100 | 102
  Probably Yes | 116 | 123
  Probably No | 18 | 25
  Definitely No | 8 | 5

5. Secondary Outcome: Treatment Choice
Description: 1 item that asked parents if their child is currently taking medication to treat their ADHD.
Time Frame: baseline survey
Population: Participants who answered the question. All 498 participants provided sufficient information for treatment choice.
Measure: Count of Participants; unit: Participants
Arm/Group | Decision Aid Arm | Control Arm
Number analyzed (Participants) | 242 | 256
Participants
  taking medication | 151 | 146
  not taking medication | 91 | 110

6. Secondary Outcome: National Initiative for Children's Healthcare Quality (NICHQ) Vanderbilt Assessment Performance Sub-scale
Description: 8 items that ask parents to rate their child's performance in school overall, in individual subjects such as reading, relationships with others such as parents and peers, and their participation in organized activities. There were 5 response options: Excellent, above average, average, somewhat of a problem, and problematic. Total scores range from 8 to 40 with higher scores indicating more problematic behavior
Time Frame: baseline survey
Population: Participants provided sufficient information to calculate a total score. Only 483/498 participants provided sufficient information
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Decision Aid Arm | Control Arm
Number analyzed (Participants) | 235 | 248
score on a scale | 22.46 (6.38) | 21.07 (6.26)

7. Secondary Outcome: Adapted Controlled Preference Scale
Description: Single item asking the parent who made the ultimate decision. The categorical response options are 1) the parent made the decision, 2)the child's provider made the decision, 3) both parent and provider made the decision together, or 4) the decision as made by someone else
Time Frame: baseline survey
Population: Participants who answered the single-item question. Only 497/498 participants provided sufficient information.
Measure: Count of Participants; unit: Participants
Arm/Group | Decision Aid Arm | Control Arm
Number analyzed (Participants) | 241 | 256
Participants
  Mainly you | 109 | 119
  Mainly your child's healthcare provider | 22 | 27
  You and the provider made the decision together | 108 | 110
  Mainly someone else | 2 | 0

8. Secondary Outcome: Shared Decision Making Process Measure Retest
Description: The Shared Decision Making Process is a short patient-reported survey that measures the amount of shared decision making that occurs in an interaction. Scores range from 0-4 where higher values indicate a better shared decision making process occurred.
Time Frame: 2 weeks after completing the baseline survey
Population: A subset of participants who completed the baseline survey were re-contacted approximately 2 weeks post baseline survey for a retest. Participants who completed the retest survey and provided enough information to calculate the shared decision making process score were part of this analysis. 208/215 provided both consistent and sufficient information.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Decision Aid Arm | Control Arm
Number analyzed (Participants) | 98 | 110
score on a scale | 2.84 (1.01) | 2.60 (1.02)

9. Other Pre Specified Outcome: Adherence
Description: 1 item measure of adherence to medication for sample of participants who indicated their child was taking medicine. The question asked "in the last 30 days, how often did your child take their ADHD medicine in the way they were supposed to?"
Time Frame: baseline survey
Population: only parents who stated their child was currently taking medicine was included in this analysis. 297 parents said their child was taking medicine, and 290/297 provided information on adherence
Measure: Count of Participants; unit: Participants
Arm/Group | Decision Aid Arm | Control Arm
Number analyzed (Participants) | 149 | 141
Participants
  Never | 5 | 5
  Rarely | 8 | 8
  Sometimes | 21 | 17
  Usually | 16 | 16
  Almost Always | 30 | 34
  Always | 69 | 61

ADVERSE EVENTS:
Time Frame: Responses were revised within 1 month of completion for evidence of adverse events
Arm/Group | Decision Aid Arm | Control Arm
All-Cause Mortality (participants affected / at risk) | 0/242 | 0/256
Serious Adverse Events (participants affected / at risk) | 0/242 | 0/256
Other Adverse Events (participants affected / at risk) | 0/242 | 0/256

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-08-10): https://cdn.clinicaltrials.gov/large-docs/86/NCT05048186/Prot_SAP_000.pdf